CLINICAL TRIAL: NCT03000920
Title: Multicenter Randomized Controlled Trial Evaluating the Effectiveness and Cost-effectiveness of the Use of Short Message Service (SMS) in the Screening Invitation Strategy for Breast Cancer.
Brief Title: Evaluation of the Short Message Service Effectiveness in the Screening Invitation Strategy for Breast Cancer (USIMaPI)
Acronym: USIMaPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: INCA15-KH/USIMaPI
Record Dates: First submitted 2016-12-12; First posted 2016-12-22 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
Keywords: short message service (SMS); screening; cost-effectiveness
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1_Control (No Intervention): Classic screening invitation strategy with at least an invitation mail and then one or two reminder by mail if necessary.
- 2_SMS Reminder 1 (Experimental): Invitation by mail then reminder 1 by SMS if necessary then reminder 2 by mail if necessary
  Interventions: Other: SMS Reminder 1
- 3_SMS before invitation (Experimental): One SMS a few days before the Invitation by mail and then one or two reminder(s) by mail if necessary.
  Interventions: Other: SMS before invitation
- 4_SMS before invitation + SMS Reminder 1 (Experimental): One SMS a few days before the Invitation by mail then reminder 1 by SMS if necessary then reminder 2 by mail if necessary
  Interventions: Other: SMS before invitation; Other: SMS Reminder 1

INTERVENTIONS:
Other: SMS before invitation — A couple of days before the invitation letter, an SMS will be sent to announce the arrival of the invitation letter to the mammogram
  Arms: 3_SMS before invitation; 4_SMS before invitation + SMS Reminder 1
Other: SMS Reminder 1 — If it is necessary for the women to have a reminder 1, the usual mail will be replaced by an SMS.
  Arms: 2_SMS Reminder 1; 4_SMS before invitation + SMS Reminder 1

SUMMARY:
Each year in France, breast cancer affects about 48,000 women and is the first cause of cancer death in women with 11,900 deaths estimated.

Since 2004, there is a national organized breast cancer screening (OBCS) programme for asymptomatic women aged 50-74 and with a medium-risk. Every two years, the local cancer screening department sends a personalized invitation mail to eligible women to perform a mammogram and a breast clinical examination. One to two reminder mails are sent to women who have not done the screening after an initial invitation. Despite this programme, almost 47% of women in France do not participate to organized breast cancer screening.

The Short Message Service (SMS) is an innovative communication tool in the field of health, immediate, reliable delivery, low cost and ecological. The use of SMS could be an innovative, low-cost, personalized and ecological way to support the OBCS invitation strategy.

The overall objective of this study is to preserve or even better increase participation in organized breast cancer screening while decreasing the associated costs by including SMS in our screening invitation procedure.

Two SMS interventions will be tested which will correspond to different phases of the OBCS invitation procedure. This sequence of interventions leads us to perform three interlinked trials: a trial of superiority for the first phase (intervention 1: sending an SMS a few days before the initial mail invitation), then two non-inferiority trials for the second phase ( two trials=one for each context of phase 1 _ intervention 2: sending an SMS in place of the first postal reminder).

DETAILED DESCRIPTION:
Each year in France, breast cancer affects about 48,000 women and is the first cause of cancer death in women with 11,900 deaths estimated.

Since 2004, there is a national organized breast cancer screening (OBCS) programme for asymptomatic women aged 50-74 and with a medium-risk. Every two years, the local cancer screening department sends a personalized invitation mail to eligible women to perform a mammogram and a breast clinical examination. One to two reminder mails are sent to women who have not done the screening after an initial invitation. Despite this programme, almost 47% of women in France do not participate to organized breast cancer screening.

The Short Message Service (SMS) is an innovative communication tool in the field of health, immediate, reliable delivery, low cost and ecological. The use of SMS could be an innovative, low-cost, personalized and ecological way to support the OBCS invitation strategy.

In databases, there is currently about 10 to 15% of the women with a mobile phone number registered in the target population.

This project will be carried out throughout the Region "Centre-Val de Loire" with six local cancer screening departments The overall objective of this study is to preserve or even better increase participation in organized breast cancer screening while decreasing the associated costs by including SMS in our screening invitation procedure.

Two SMS interventions will be tested which will correspond to different phases of the OBCS invitation procedure. This sequence of interventions leads us to perform three interlinked trials: a trial of superiority for the first phase (intervention 1: sending an SMS a few days before the initial mail invitation), then two non-inferiority trials for the second phase (intervention 2: sending an SMS in place of the first postal reminder).

Justification of methodological choices

1. st phase: Addition of the intervention "sending an SMS" (and the associated cost) to what is currently done (versus classical intervention). To be of interest, the tested intervention, the sending of an SMS few days before the initial mail invitation, should allow to significantly increase participation in OBCS (here superiority trial).
2. nd phase: This phase will involve women who have had or not the phase 1 intervention and who have not yet participated to the OBCS. Since the contexts in phase 1 are different, a trial for each one must be carry out. In this second phase, the conventional intervention (sending reminder mail 1) will be compare to a cheaper one (sending reminder 1 by SMS). The new strategy will prove interesting if it is not inferior in terms of participation to the OBCS. The analysis of this non-inferiority will be carried out for each context of phase 1 (invitation mail alone OR SMS then invitation mail).

The 4 groups of the study are the followings:

* Group 1 (usual procedure): at least an invitation mail and then one or two reminder by mail if necessary.
* Group 2 : Invitation by mail then reminder 1 by SMS if necessary then reminder 2 by mail if necessary
* Group 3 : One SMS a few days before the Invitation by mail and then one or two reminder(s) by mail if necessary
* Group 4 : One SMS a few days before the Invitation by mail then reminder 1 by SMS if necessary then reminder 2 by mail if necessary

ELIGIBILITY:
Inclusion Criteria:

* eligible to the organized breast cancer screening
* residing in the region of Centre-Val de Loire (France)
* Phone number registered in data bases of one of the 6 local cancer screening departments of the region of Centre-Val de Loire (France)

Exclusion Criteria:

* none

Ages: 50 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12000 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Phase 1: Compare the participation rates in organized breast cancer screening (and the cost by screened woman) in response to a strategy of sending an SMS before the invitation letter (vs sending the invitation letter alone = usual strategy). | Before the sending time of the reminder 1 (letter or SMS) : from 3 months to 8 months after the invitation letter depending to periods of the concerned local cancer screening department
  For this first phase, the study aims to demonstrate that the addition of the SMS is superior in terms of participation and participation costs.
Phase 2: Compare participation rates in organized breast cancer screening (and the cost by screened woman) in response to a strategy of replacing the reminder 1 by mail with a reminder 1 by SMS ( reminder 1 mail = usual strategy). | Before the sending time of the reminder 2 : from 3 months to 6 months after the reminder 1 depending to periods of the concerned local cancer screening department
  For this second phase, the study aims to demonstrate the non-inferiority of the strategy including the SMS in terms of participation and cost-participation according to the two contexts:
  * women who have already received an invitation letter alone.
  * women who have already received one SMS and the invitation mail.

CONTACTS AND LOCATIONS:
Overall Officials: ken HAGUENOER, Dr, Principal Investigator — Centre de Coordination des Dépistages des Cancers, CHRU de Tours; Somany SENGCHANH, Dr, Principal Investigator — Centre de Coordination des Dépistages des Cancers, CHRU de Tours; Julie Boyard, Principal Investigator — Centre de Coordination des Dépistages des Cancers, CHRU de Tours
Locations (4):
- France (4):
  - ADOC41, Blois
  - ADOC28, Chartres
  - CREDEP, Châteauroux
  - CCDC, Tours

IPD SHARING:
Plan to Share IPD: No